CLINICAL TRIAL: NCT04041401
Title: A Paediatric Intensive Care Unit (PICU) 'Storybooks' Intervention for Children and Their Caregivers: a Case-series Feasibility Study
Brief Title: The Experiences of Children and Caregivers Given PICU Storybooks
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SPON 2018 021 FHMS
Record Dates: First submitted 2019-06-05; First posted 2019-08-01 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: PTSD; Critical Illness; Depression; Anxiety; Quality of Life
Keywords: paediatric intensive care unit; intervention; PTSD; storybook; Narrative; Feasibility; Case-series
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Critical Illness; Depression; Anxiety Disorders; Narration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and their Caregivers: Children following discharge from PICU and their caregivers receiving a storybook intervention.
  Interventions: Other: PICU storybook

INTERVENTIONS:
Other: PICU storybook — Narrative and developmentally appropriate intervention

SUMMARY:
1. To assess the acceptability and feasibility of a study design aimed at evaluating the efficacy of a newly developed intervention for children and their caregivers following discharge from PICU
2. To assess the acceptability of the newly developed 'storybook intervention'

DETAILED DESCRIPTION:
Admission to a Paediatric Intensive Care Unit (PICU) can be extremely stressful for patients and their caregivers. Both are at heightened risk of psychological distress, including post-traumatic stress symptoms (PTSS), which sometimes persist for months or years post-discharge. Unfortunately, few post-PICU psychological interventions have been studied. Documented challenges in PICU research (e.g. low recruitment rates) means feasibility issues require investigation before investing resources in intervention trials.

In adult intensive-care, diaries are used to help patients and families undergo key processes that underpin therapies to reduce PTSS: talking about and understanding their experiences. In the only published study exploring paediatric ICU diaries, families gave positive feedback, but their clinical effectiveness has not yet been evaluated. Further, it is hypothesised that formatting diaries as 'storybooks' is more adaptable to the developmental variation of the paediatric population.

Using a case-series design, this research aims to establish the feasibility of recruiting to a study evaluating PICU storybooks. It will explore the acceptability of research tasks to families, the utility and sensitivity of psychometric measures, plus how storybooks are used and perceived in supporting psychological recovery. It is anticipated that the findings will directly inform the planning of a larger scale evaluation study, and adaptations to the intervention. The hope is this will lead to improved support for families leaving PICU.

Pairs of caregivers and their children aged 3-15 will be recruited upon discharge from a PICU and will receive an individualised, developmentally-appropriate storybook about their PICU experiences. At discharge, and one, three and six months post-discharge, caregivers and children aged 8+ will complete questionnaires about psychological distress symptoms (depression, anxiety and PTSS) and their impact on functioning. Participants will be asked to keep a brief log of their storybook use and will be interviewed about their experience of the intervention and research procedures at three and six months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Parent-child dyads where the child has been admitted to the St Georges Hospital PICU during the recruitment phase.
2. At time of discharge, the parent is at least 18 years old, and the child is between 3 and 15 years old with an assumed cognitive ability of at least 3 years.
3. Child's admission was at least 24 hours in duration.

Exclusion Criteria:

1. Parent-child dyads that do not meet all inclusion criteria above, or;
2. The child's admission was due to a non-accidental injury or they are known to be the subject of safeguarding concerns within their family;
3. Either the parent or child has a severe visual impairment, or the parent is unable to read.
4. The child is 'Looked after'/in foster care.
5. The child is discharged from PICU to end of life care.
6. Either the parent or child is participating in other intervention research for PICU survivors, is in receipt of psychological therapy in relation to the admission, or has already received a storybook about this most recent PICU admission.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients and their caregivers admitted to the PICU at St George's Hospital PICU.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rate | 6 months
  Percentage of participants approached, recruited and retained.
Questionnaire completion rate | 6 months
  Percentage of questionnaires administered that were completed.
Success rate of intervention delivery within 4-6 weeks post-discharge | 6 months
  Proportion of storybooks given to family within 6 weeks
Acceptability of intervention and research participation: qualitative interview | 3 months
  Child and parent reported qualitative interview data regarding acceptability of intervention and research design in the first three months.
Acceptability of intervention and research participation: qualitative interview | 6 months
  Child and parent reported qualitative interview data regarding acceptability of intervention and research design over six months.

SECONDARY OUTCOMES:
Post-traumatic Adjustment Screen (parent participants) | 24 hours
  This is a brief measure consisting of 10 items that ask parents to rate the extent to which they experienced factors relating to before, during or after their child's intensive care unit stay. Each item is rated on a 5 point scale, from 0= not at all to 4=totally. Scores are summed to provide a total (0- 40), with totals above 16 indicating risk of post-traumatic stress.
Work and Social Adjustment scale (parent participants; change being assessed) | 24 hours, 1 month, 3 months and 6 months
  This is a five-item measure assessing functional impairment in relation to work, home management, social leisure activities, private leisure activities, and family and relationships. Each item is rated on a nine-point scale ranging from 0 (no impairment) to 8 (severe impairment) and all items scores are added together to give a total score indicating mild (0-9), moderate (10-19) or severe (20-40) impairment.
Paediatric Quality of Life (PedsQL) (child participants; change being assessed) | 24 hours, 1 month, 3 months and 6 months
  The PedsQL is a 23-item generic measure of health-related quality of life divided into four dimensions (Physical, Emotional, Social, School) designed for 2-18 year olds. It is available in four separate versions for ages 2-4, 5-7, 8-12 and 12-18 year olds (self-report versions available for children 8 years and above). Each item is rated on a 5-pint scale from 0=never, to 4=almost always, where 0= a score of 100, 1= score of 75, 2=score of 50, 3=score of 25 and 4= score of 0. Scores from different items can be summed to compute two Summary Scores (the Psychosocial Health Summary Score and the Physical Health Summary Score), or all can be summed to provide a total score. Higher scores indicate better health related quality of life.
Strength and Difficulties Questionnaire (SDQ) (child participants; change being assessed) | 24 hours, 1 month, 3 months and 6 months
  The SDQ comprises of 25 questions on psychological attributes, divided into five 5-item symptom subscales: Conduct Problems, Peer relationships, Emotional Symptoms, Hyperactivity-Inattention, and Prosocial Behaviour. Items are rated on 3-point scale (0= not true, 1= somewhat true, 2= certainly true) and summed to provide total scores for each scale.
The Hospital Anxiety and Depression Scale (HADS) (for parent participants; change being assessed) | 24 hours, 1 month, 3 months and 6 months
  This is a self-report scale containing two 7- item Likert subscales to assess the presence of symptoms of anxiety and depression. Items are rated on a scale from 0-3, with higher scores indicating greater symptom severity. Items are combined and summed to give a total score for anxiety and a total score for depression symptoms.
The PTSD (post traumatic stress disorder) Checklist for DSM (diagnostic statistical manual) 5 (PCL5) (for parent participants; change being assessed) | 1 month, 3 months and 6 months
  This is a 20-item self-report measure in which participants rate how much they are bothered by symptoms of PTSD on a 5-point scale (0 = "Not at all" to 4 = "Extremely"). A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items, with scores of 33-80 indicating clinical levels of symptoms.
The Child revised Impact of Events Scale - 8 (CRIES-8) (For child participants; change being assessed) | 1 month, 3 months and 6 months
  This is an 8-item self report measure in which participants rate how much they experience symptoms of PTSD on a 4-point scale (0= not at all, 1=rarely, 3=sometimes, 5=often). Scores are added together to give a total score (0-40), with scores over 17 suggestive of clinical levels of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ellie Atkins, Principal Investigator — St George's Hospital Paediatric Psychology
Locations (1):
- St George's Hospital, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided